CLINICAL TRIAL: NCT01929447
Title: A Prospective, Comparative Study to Evaluate the Watch-PAT200 (WP200) With the Unified Probe (WP200U) Compared to the Currently Used Configuration of WP200 With the Nonin Oximetry Module
Brief Title: Evaluation of WP200 With the Unified Probe (WP200U)
Status: Completed | Type: Observational
Sponsor: Itamar-Medical, Israel (Industry)
Responsible Party: Sponsor
Other Study IDs: Carmel-002
Record Dates: First submitted 2013-08-20; First posted 2013-08-28 (Estimated); Last update posted 2014-09-19 (Estimated); Status verified 2014-09

CONDITIONS: Sleep Disorders
Keywords: sleep disorders; sleep apnea; ambulatory device; WatchPAT
MeSH Terms: conditions — Sleep Wake Disorders; Sleep Apnea Syndromes

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The prevalence of OSAS is estimated at 2% and 4% for adult women and men respectively, most of whom are undiagnosed and untreated. The severity of the disorder is expressed by the Apnea Hypopnea Index (AHI) which is the number of Apnea/Hypopnea episodes per hours of actual sleep and the Respiratory Disturbances Index (RDI) which is an extended index incorporating in addition to the previous episodes also respiratory effort related arousal episodes. The high cost of in-lab full night PSG, together with long waiting lists for sleep studies, have led to the development of a variety of ambulatory sleep study systems.

The primary objective of the study is to evaluate the newly developed WP200 with the unified probe (WP200U) compared to the currently used configuration of WP200 that uses an incorporated Nonin oximetry module in the sleep lab or in the home sleep environment.

ELIGIBILITY:
Inclusion Criteria:

* Age between 5-90
* Subjects that are able to read understand and sign the informed consent form of the study or by parents of subjects that are less than 18 years of age that are either referred or volunteering to undergo an overnight sleep study in the clinical sleep laboratory or at home

Exclusion Criteria:

* Permanent pacemaker.
* Severe lung disease.
* Severe peripheral neuropathy.
* Finger deformity that precludes adequate sensor appliance.
* Using one of the following medications: short/Long acting nitrates (less than 3 hours before the sleep study) or alpha-adrenergic receptor blockers (less than 24 hours before the sleep study).

Ages: 5 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Subjects, adults and children, with suspected sleep disorders who are referred to a sleep study and are willing to participate in this clinical study.
  Additional non selective volunteers who are willing to participate in this clinical study and consent to undergo an overnight sleep study at their home.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2013-10; Primary Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Sleep respiratory parameters | 3 years
  pRDI, pAHI, ODI

CONTACTS AND LOCATIONS:
Locations (1):
- Carmel Medical Center, Haifa, Israel